CLINICAL TRIAL: NCT00844558
Title: Optimizing Mobility in Older Adults With Knee Osteoarthritis
Brief Title: Mobility Optimization Through Velocity Exercise
Acronym: MOVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Neil A Segal, Associate Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 200807706; K23AG030945-01 (NIH)
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Results first posted 2016-06-06 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-05

CONDITIONS: Knee Osteoarthritis
Keywords: osteoarthritis; knee pain; gait training; power training; rehabilitation; physical therapy
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gait Training (Experimental): Gait Training Intervention Group Participants
  Interventions: Other: Gait Training
- Control (Placebo Comparator): Gait Training Control Group Participants
  Interventions: Other: Control

INTERVENTIONS:
Other: Gait Training — Gait training with a physical therapist 2/week for the first 3 months followed by 1/week for the following 3 months
  Arms: Gait Training
Other: Control — There is no intervention associated with this arm of the study
  Arms: Control

SUMMARY:
Knee Osteoarthritis (OA) accounts for a significant proportion of mobility limitations and is one of the most disabling problems facing the growing population of older adults. The purpose of this research is to reduce disablement of older adults with symptomatic knee osteoarthritis.

DETAILED DESCRIPTION:
The long-term objective of this research is to reduce disablement of older adults with knee osteoarthritis (OA). This will be accomplished through assessing changes in functional limitations (standing and walking) that occur with 2 mobility-specific interventions. The principle of specificity of training indicates that exercises that closely approximate the goal functional activity are most effective in improving physical performance during that activity. However, there is uncertainty whether intervening to increase muscle power or to improve gait mechanics would be most effective for optimizing mobility in older adults with knee OA. Although gait training may be most specific for improving gait, this approach currently requires supervised physical therapy and expensive equipment. In contrast, power training may be less costly and more convenient if conducted at home. To optimize mobility in older adults with symptomatic knee OA, there is a need to study each of these mobility-specific interventions in a randomized controlled trial (RCT). Successful completion of this trial will inform rehabilitation for maintaining or improving mobility as well as explore the mechanism of effect.

Specific Aim 1: Assess the efficacy of two innovative interventions for improving mobility limitations, disability and quality of life in older adults with symptomatic knee OA.

Primary Hypothesis: For older adults with symptomatic knee OA, in comparison with usual care (control group), a 3-month a) patient-specific gait training intervention and b) mobility-specific power training intervention will reduce lower limb mobility limitations assessed using the Function component of the Late Life Function and Disability Index (LLFDI-Function).

Hypothesis 2: Improved mobility will be maintained at 6 and 12-month follow-up (3 and 9 months following transitioning to home-based training) for each of the 2 intervention groups who receive the combination of the home-based intervention and encouragement to continue participation.

Hypothesis 3: In comparison to baseline measures, at 3, 6, and 12-month follow-up, each of the 2 intervention groups will demonstrate improvements in a) disability (LDCW), b) quality of life assessed using the Knee Osteoarthritis Outcome Score questionnaire Quality of Life component(KOOS Knee QOL), and c) knee OA specific outcome scores using the pain subscale component of KOOS.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 or older
* Symptomatic knee osteoarthritis (knee osteoarthritis diagnosed by x-ray and frequent knee symptoms)

Exclusion Criteria:

* bilateral knee replacement
* acute or terminal illness
* unstable cardiovascular condition or other medical conditions that may impair ability to participate such as pulmonary disease requiring use of supplement oxygen, or current medical condition that affects walking, or lower limb musculoskeletal surgery in the past 6 months

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2008-08; Primary Completion 2010-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil A Segal, MD, MS, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Gait: Gait Training Arm
  Gait Training: Gait training with a physical therapist 2/week for the first 3 months followed by 1/week for the following 3 months
- Control: Control Group
  Control: There is no intervention associated with this arm of the study
Period: Overall Study
Arm/Group | Gait | Control
Started | 36 (* Received allocated intervention (n=33) * Did not receive allocated intervention (n=3)) | 22 (* Received allocated intervention (n=21) * Did not receive allocated intervention (n=1))
Received Allocated Intervention | 33 | 21
3 Month Visit | 29 (Discontinued intervention (n=4)) | 19 (* Lost to follow-up (n=1) * Discontinued Intervention (n=1))
6 Month Visit | 28 (Discontinued intervention (n=1)) | 18 (-Discontinued intervention (n=1))
12 Month Visit | 24 (Discontinued intervention (n=4)) | 18 (-Discontinued intervention (n=0))
Completed | 24 | 18
Not Completed | 12 | 4
Not completed — Withdrawal by Subject | 9 | 2
Not completed — Death | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: The objective of this study was to determine whether individualized gait training is more effective than usual care for reducing mobility disability and pain in individuals with symptomatic knee osteoarthritis.
Groups:
- Gait: The gait participants were randomized and attended 24 biweekly 45-minute sessions directed by a physical therapist, which were composed of guided strategies to optimize knee movements during treadmill walking, using computerized motion analysis with visual biofeedback.
- Control: The control participants received their usual care for symptomatic knee osteoarthritis (OA) through their usual healthcare providers and were not asked to make changes to their lifestyle.Usual care for these subjects may have included a yearly visit with their physician, use of pain medications for knee symptoms, knee surgery, and/or physical therapy.
- Total: Total of all reporting groups
Arm/Group | Gait | Control | Total
Number analyzed (Participants) | 36 | 22 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (7.3) | 69.6 (6.4) | 69.3 (7.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 10 | 32
  Male | 14 | 12 | 26
Region of Enrollment [Number; unit: participants]
  United States | 36 | 22 | 58

OUTCOME MEASURES:

1. Primary Outcome: Change in Basic Lower Limb Function (Late Life Function Index) Late Life Function and Disability Instrument
Description: This is a questionnaire that evaluates self-reported difficulty in a person's ability to do discrete actions or activities primarily involving standing, stooping and fundamental walking activities without the help of others. Factors that may influence difficulty in task performance include pain, fatigue, fear, weakness, soreness, ailments, health conditions and disabilities.
  Scored from 14 to 70 with scores approaching 70 signifying high levels in ability to perform activities primarily involving standing, stooping, and fundamental walking (without assistance), and scores approaching 14 signifying low levels in ability to perform activities primarily involving standing, stooping, and fundamental walking (without assistance).
Time Frame: 0,3,6, and 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Gait; Control Group: No adverse events
Arm/Group | Gait | Control Group
Number analyzed (Participants) | 29 | 19
units on a scale
  Change from baseline to month 3 | 3.3 [1.1 to 5.5] | -1.0 [-3.7 to 1.7]
  Change from baseline to month 6 | 3.1 [0.5 to 5.7] | 0.8 [-2.3 to 4.0]
  Change from baseline to month 12 | 3.9 [-1.3 to 9.1] | 2.9 [-3.7 to 9.5]

2. Secondary Outcome: Change in Knee Osteoarthritis Injury and Outcome Scale (KOOS) Pain
Description: This is a 42-item self-administered questionnaire that covers five patient-relevant dimensions, including pain and knee-related symptoms. This instrument has been found to be a reliable and responsive measure in older adults with knee OA as well as sensitive to changes in pain and knee-related symptoms over 6- and 12-mo periods.
  Scored from 0 to 100 with 100 indicating no pain.
Time Frame: 0,3,6 and 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Gait | Control
Number analyzed (Participants) | 29 | 19
units on a scale
  Change from baseline to month 3 | 8.2 [2.8 to 13.5] | 1.1 [-5.5 to 7.7]
  Change from baseline to month 6 | 5.4 [0.1 to 10.7] | 1.7 [-4.8 to 8.2]
  Change from baseline to month 12 | 10.1 [4.4 to 15.8] | 2.8 [-4.4 to 10.1]

3. Secondary Outcome: Change in KOOS Symptoms
Description: This instrument has been found to be a reliable and responsive measure in older adults with knee OA as well as sensitive to changes in pain and knee-related symptoms over 6- and 12-mo periods.
  Scored from 0 to 100 with 100 indicating no symptoms.
Time Frame: 0,3,6 and 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Gait | Control
Number analyzed (Participants) | 29 | 19
units on a scale
  Change from baseline to month 3 | 11.5 [6.3 to 16.7] | 3.0 [-3.4 to 9.4]
  Change from baseline to month 6 | 8.1 [2.3 to 13.8] | 1.8 [-5.3 to 8.9]
  Change from baseline to month 12 | 8.5 [0.9 to 16.0] | 2.4 [-7.1 to 12.0]

4. Secondary Outcome: Change in Long Distance Corridor Walk (LDCW) Time, Secs
Description: The LDCW included both 2-min walk distance and 400-m walk time. This measure has been shown to be predictive of changes in community mobility. Per the LDCW protocol, for participants unable to walk 400 m, gait speed was estimated from the 2-min walk distance, so that all participant data were on the same scale.
Time Frame: 0,3,6 and 12 months
Measure: Mean (95% Confidence Interval); unit: seconds
Groups:
- Control: No adverse events
Arm/Group | Gait | Control
Number analyzed (Participants) | 29 | 19
seconds
  Change from baseline to month 3 | 11.5 [6.3 to 16.7] | 3.0 [-3.4 to 9.4]
  Change from baseline to month 6 | 8.1 [2.3 to 13.8] | 1.8 [-5.3 to 8.9]
  Change from baseline to month 12 | 8.5 [0.9 to 16.0] | 2.4 [-7.1 to 12.0]

5. Secondary Outcome: Change in Stair Climb Time, Secs
Description: Functional limitations specific to ascending stairs were assessed with a times stair climb, using a standard eight-stair flight (stair height = 19 cm)
Time Frame: 0,3,6, and 12 months
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Gait Training | Control
Number analyzed (Participants) | 29 | 19
seconds
  Change from baseline to month 3 | 0.2 [-0.5 to 0.9] | 0.0 [-0.9 to 0.8]
  Change from baseline to month 6 | -0.2 [-1.3 to 1.0] | -1.4 [-2.9 to 0.0]
  Change from baseline to month 12 | -0.3 [-1.3 to 0.7] | -1.1 [-2.4 to 0.1]

6. Secondary Outcome: Change in Chair Stand Time
Description: Measured as the total time (in seconds) required to stand five times from a seated position in a standardized chair without using arms.
Time Frame: 0,3,6,and 12 months
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Gait | Control
Number analyzed (Participants) | 29 | 19
seconds
  Change from baseline to month 3 | -0.9 [-2.2 to 0.4] | -1.0 [-2.8 to 0.8]
  Change from baseline to month 6 | -1.9 [-3.5 to -0.3] | -3.0 [-5.0 to -0.9]
  Change from baseline to month 12 | -2.5 [-3.7 to -1.3] | -2.9 [-4.5 to -1.3]

ADVERSE EVENTS:
Time Frame: 1 year
Description: Clinical Data Safety Monitor reviewed adverse event reports quarterly.
Groups:
- Gait: Gait training with a physical therapist 2/week for the first 3 months followed by 1/week for the following 3 months
- Control: Usual care for symptomatic knee OA through their usual healthcare providers and were not asked to make changes in their lifestyle. Usual care may have included a yearly visit with their physician, use of pain medications for knee symptoms, knee surgery and/or physical therapy.
Arm/Group | Gait | Control
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/22
Other Adverse Events (participants affected / at risk) | 0/36 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No